CLINICAL TRIAL: NCT00410566
Title: A Phase I, Single-Center, Single Dose, Dose Escalation Study of Recombinant Human Acid Sphingomyelinase (rhASM) in Adults With Acid Sphingomyelinase Deficiency (ASMD)
Brief Title: Safety Study of rhASM Enzyme Replacement Therapy in Adults With Acid Sphingomyelinase Deficiency (Niemann-Pick Disease)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated by sponsor - Single dose safety objective achieved.
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPHINGO00605
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Acid Sphingomyelinase Deficiency; Niemann-Pick Disease
Keywords: Acid sphingomyelinase deficiency; Niemann-Pick disease; Lysosomal storage disorder; Enzyme replacement therapy; Treatment
MeSH Terms: conditions — Niemann-Pick Diseases; Lysosomal Storage Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: rhASM
- 2 (Experimental)
  Interventions: Drug: rhASM
- 3 (Experimental)
  Interventions: Drug: rhASM
- 4 (Experimental)
  Interventions: Drug: rhASM
- 5 (Experimental)
  Interventions: Drug: rhASM

INTERVENTIONS:
Drug: rhASM — Single dose of 0.03mg/kg body weight IV
  Arms: 1
Drug: rhASM — Single dose of 0.1mg/kg body weight IV
  Arms: 2
Drug: rhASM — Single dose of 0.3mg/kg body weight IV
  Arms: 3
Drug: rhASM — Single dose of 0.6mg/kg body weight IV
  Arms: 4
Drug: rhASM — Single dose of 1.0mg/kg body weight IV
  Arms: 5

SUMMARY:
The purpose of this study is to determine the safe range of single doses of rhASM administered to adults with ASM deficiency.

DETAILED DESCRIPTION:
ASM deficiency (ASMD), also known as Niemann-Pick A and B disease, is a rare genetic disorder in which reduced activity of the lysosomal enzyme, ASM, leads to the accumulation of sphingomyelin primarily in macrophages throughout the body. This deficiency results in characteristic features such as hepatosplenomegaly, thrombocytopenia, interstitial lung disease, growth retardation, coronary artery disease, fatigue, and in severe cases, neurodegeneration with death in early childhood. There is no specific treatment for this disease. This Phase 1 safety study will seek to enroll a minimum of 12 and a maximum of 30 eligible adults patients with ASMD with each patient participating for approximately 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed, informed consent by the patient or legal guardian prior to performing any study-related procedures;
* Have ≤ 0.2 nmol/hr/mg protein ASM activity in peripheral leukocytes, as measured by the reference laboratory;
* Have a diffusing capacity (DLco) > 30% of the predicted normal value;
* Have a spleen volume ≥ 2x normal
* Female patients of childbearing potential must have a serum pregnancy test negative for β-hCG and agree to use a reliable birth control method for the duration of the study.

Exclusion Criteria:

* Is pregnant or lactating;
* Has received an investigational drug within 30 days prior to study enrollment;
* Has a medical condition, including serious intercurrent illness, active hepatitis B or C or human immunodeficiency virus (HIV) infection, cirrhosis, > stage 3 liver fibrosis, INR >1.5, platelet count < 60.0x10^3/µL, significant cardiac disease (e.g. pulmonary artery pressure > 40 mm Hg, moderate or severe valvular dysfunction, or < 40% left ventricular ejection fraction by echocardiography (ECHO)), or any other extenuating circumstances that may significantly interfere with study compliance including all prescribed evaluations and follow-up activities;
* Has had a major organ transplant (e.g. bone marrow or liver);
* Has had a total splenectomy;
* Has an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value >250 IU/L or a total bilirubin >3.6 mg/dL;
* Is unwilling or unable to avoid the use of alcohol, medications that may decrease rhASM activity, medications or herbal supplements that may cause or prolong bleeding, and the use of medications or herbal supplements with potential hepatoxicity within 14 days prior to and 28 days afte the rhASM infusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-12; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Safety assessments via physical exam,AE reporting,telemetry heartrate monitoring,ECG,ECHO,clinical lab evaluations,liver and adrenal function tests,cytokine testing,adrenal hormone levels,lipid profile,chest Xrays,liver biopsies,MRI of internal | Pre-, During-, and Post-infusion (up to 72 hrs); 14 day and 28 day follow-up visit
Immune Response Measure | Pre-infusion and final visit (Day 28)

SECONDARY OUTCOMES:
PK measurements | Pre- and Post-infusion up to 72 hrs.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- New York, New York, United States